CLINICAL TRIAL: NCT04188600
Title: National, Multicentric, Randomized, Single-blind, Active-controlled Phase III Clinical Trial to Evaluate the Efficacy and Safety of Libicare® in Women With Low Arousal and Sexual Desire Levels
Brief Title: Study to Evaluate the Effectiveness and Safety of Libicare® in Women With Low Arousal and Sexual Desire Levels
Acronym: VITAL
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision
Sponsor: Procare Health Iberia S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VITAL STUDY
Record Dates: First submitted 2019-11-27; First posted 2019-12-06 (Actual); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Female Sexual Interest/Arousal Disorder

STUDY DESIGN:
Intervention Model Description: The selected patients will be randomly distributed in one of the two arms (Libicare® / active-control), in a 2:1 ratio according to a randomization list. The kits containing the study treatment (Libicare®) and the active-control will be numbered with a randomization code according to this unique list and will be distributed to the consultations.
  Patients will not know the treatment and only the researchers and team investigator assigned to the study will know the treatment assigned.
  A second randomization list (ratio 1:1) will be generated for Libicare® responding patients, at 12 weeks in order to assign two sub-groups: continue Libicare® treatment or observation without Libicare® treatment.
Who Masked: Participant, Investigator
Masking Description: The analysis of the results will be blind for the investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- treatment group (Experimental): The treatment group will be treated with Libicare for three month (2 tablets/day). After the first three months (12 weeks) of treatment, the treatment group will be classified into two populations:
  * Responding patients: this population, defined by FSFI score > 26.55, will be randomized (1:1) into 2 groups: one of them will take Libicare® for further 12 weeks (total period on treatment: 24 weeks) and the other group will remain under observation with no treatment for further 12 weeks (total period on treatment: 12 weeks).
  * Non-responding patients: this population, defined by FSFI score ≤ 26.55, will intake Libicare® for further 12 weeks (total period on treatment: 24 weeks).
  Interventions: Dietary Supplement: Libicare
- active control group (Active Comparator): The active control group will be treated with a Selenium and vitamins B complex for three month (2tablets/day). After the first three months (12 weeks) of treatment, patients of the active-control group will cross over the treatment to Libicare® for three months (12 weeks)
  Interventions: Dietary Supplement: Libicare; Dietary Supplement: active control

INTERVENTIONS:
Dietary Supplement: Libicare — The main ingredients of Libicare® are:
  * Trigonella Foenum-graecum (Trigonella)
  * Tribulus Terrestris (Tribulus)
  * Turnera Diffusa (Damiana)
Dietary Supplement: active control — Selenium and vitamins B complex
  Arms: active control group

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Libicare® in the sexual desire and arousal at 12 weeks in peri or postmenopausal women aged between 40 and 60 years old with low sexual desire and arousal compared with active control.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the effectiveness of Libicare® in the sexual desire and arousal at 12 weeks in peri or postmenopausal women aged between 40 and 60 years old with low sexual desire and arousal compared with active control.

Despite current consensus in the literature that Female Sexual Dysfunction can manifest at any age in a woman´s life, researchers as Sarrel documented that during menopause, up to 40% of women are experiencing a decrease in their sexual libido. The common assumption is that the menopause contributes to a drop of the sexual desire probably as a result of low production of hormones from ovaries, at the same time will reduce the estrogen and testosterone. This reduction starts to be reduced in the thirties and continues to reduce progressively at a constant rate reaching of about 50% of their initial highest levels by the time they reach menopause. Other hormones could be involved as Sex hormone-binding globulin (SHBG) or dehydroepiandrosterone (DHEA), both are related with testosterone levels.

Libicare® is a dietary supplement whose ingredients could have positive effects on the improvement of sexual function in women with low desire and arousal levels.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged between 40 and 60 years old.
2. Healthy peri or postmenopausal women.
3. Body Mass Index (BMI) between 18,5-29,9.
4. Female with low sexual desire and low arousal with a score ≤26.55 on the questionnaire Female Sexual Function Index (FSFI) .
5. Patients who signed the Informed Consent Form.

Exclusion Criteria:

1. Female with uncontrolled thyroid function.
2. Female with severe genital pain (vaginism, stopping intercourse because of severe pain).
3. Female diagnosed with primary female orgasmic disorder.
4. No coital intercourse a month.
5. Lack of steady sexual partner.
6. Suffering from any serious medical condition (any disease which may force the participant to use drug during the study).
7. Suffering from major depression disorder or other psychiatric disorders.
8. Women on anticoagulant treatment.

Min Age: 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Peri or postmenopausal women older 45 years with low sexual desire and arousal
Enrollment: 0 (Actual)
Dates: Start 2019-11-14 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Evolution of sexual desire and arousal | 12 weeks
  The evolution of the composite score from sexual desire and arousal obtained using FSFI (Female Sexual Function Index) questionnaire. It has 19 questions with six domains included desire, arousal, lubrication, orgasm, satisfaction and pain, and a general score in which higher scores reflected better sexual activity.

SECONDARY OUTCOMES:
The evolution of the composite score from sexual desire and arousal | at 6 and 24 weeks
  The evolution of the composite score from sexual desire and arousal obtained using FSFI (Female Sexual Function Index) questionnaire. It has 19 questions with six domains included desire, arousal, lubrication, orgasm, satisfaction and pain, and a general score in which higher scores reflected better sexual activity.
The evolution of the FSFI questionnaire total score | at 6, 12 and 24 weeks
  The evolution of the FSFI (Female Sexual Function Index) questionnaire total score. Composite score from sexual desire and arousal domains will be calculed as the sum of desire items (2 questions) and arousal items (4 questions). Higher scores reflected better sexual activity.
The evolution of other each sexual FSFI domain score | at 6, 12 and 24 weeks
  The evolution of other each sexual FSFI domain score (Female Sexual Function Index) It contains 2 questions of desire domain and 4 questions of arousal domain. Higher scores reflected better sexual activity.
To evaluate the hormonal levels (free testosterone and SHBG) | at 6, 12 and 24 weeks
  changes in hormonals levels
The evolution of the vitality status obtained using the Subjective Vitality Scale questionnaire | at 12 and 24 weeks
  The evolution of the vitality scale (an 7-point Likert Scale) contains 7 items. Higher scores reflected better vitality status.
The improvement in the Quality of life of women by EQ-5D-5L questionnaire | at 12 and 24 weeks
  The improvement in the Quality of life of women by EQ-5D-5L (European Quality of Life-5 Dimensions) questionnaire. It comprises the same 5 dimensions (mobility, self care, usual activities, pain/discomfort, and anxiety/depression). Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems, and extreme problems. The result is in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.
Clinical satisfaction of the women with the treatment, using a Likert-type scale | at 6, 12 and 24 weeks
  Clinical satisfaction of the women with the treatment, using a Likert-type scale of 7 points (from 1 = Very satisfied to 7 = Very dissatisfied)
The improvement of is frequency of intercourse and non-intercourse activity (total and satisfying events), number of orgasms using the SAL© | at 6, 12 and 24 weeks
  The improvement of is frequency of intercourse and non-intercourse activity (total and satisfying events), number of orgasms using the SAL© ((Sexual Activity Log©). It is a weekly diary that it measures frequency of intercourse and non-intercourse activity (total and satisfying events), number of orgasms.
The evaluation of the degree of therapeutic compliance | at 6, 12 and 24 weeks
  The evaluation of the degree of therapeutic compliance throught Likert Scale of 5 points (from 1 = Very satisfied to 5 = Very dissatisfied) will be analysed by means of percentage.
Adverse events and adverse drug reactions | at 6, 12 and 24 weeks.
  To evaluate the safety of libicare measuring the incidence and duration of adverse events and adverse drug reactions.
Weight, height and BMI | at baseline, 6, 12 and 24 weeks
  Safety endpoint for evaluating weigh and BMI (body mass index) changes.

CONTACTS AND LOCATIONS:
Overall Officials: Josep Combalia, MD, Study Director — Procare health Iberia
Locations (1):
- Procare Health Iberia, Castelldefels, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Rao A, Steels E, Beccaria G, Inder WJ, Vitetta L. Influence of a Specialized Trigonella foenum-graecum Seed Extract (Libifem), on Testosterone, Estradiol and Sexual Function in Healthy Menstruating Women, a Randomised Placebo Controlled Study. Phytother Res. 2015 Aug;29(8):1123-30. doi: 10.1002/ptr.5355. Epub 2015 Apr 24. PMID 25914334
- [Result] Akhtari E, Raisi F, Keshavarz M, Hosseini H, Sohrabvand F, Bioos S, Kamalinejad M, Ghobadi A. Tribulus terrestris for treatment of sexual dysfunction in women: randomized double-blind placebo - controlled study. Daru. 2014 Apr 28;22(1):40. doi: 10.1186/2008-2231-22-40. PMID 24773615
- [Result] Zhao J, Dasmahapatra AK, Khan SI, Khan IA. Anti-aromatase activity of the constituents from damiana (Turnera diffusa). J Ethnopharmacol. 2008 Dec 8;120(3):387-93. doi: 10.1016/j.jep.2008.09.016. Epub 2008 Sep 26. PMID 18948180